Apnimed, Inc.

Protocol: SEED

Clinical Study Protocol

# **Title Page**

Protocol Title: Open-Label 4-Period Dose-Escalation Safety and Efficacy Study of AD313 in

Participants With Obstructive Sleep Apnea

**Protocol Name: SEED** 

**Version Number:** 1.0

**Compound Number:** AD313

**Short Title:** <u>S</u>tudy for <u>E</u>fficacy and Dose <u>E</u>scalation of <u>D</u>ronabinol + Atomoxetine (SEED)

**Sponsor Name and Legal Registered Address:** 

Apnimed, Inc.

20 Holyoke Street

Cambridge, MA 02138

**Approval Date:** 25 June 2021

Date and Version of Previous Protocol: n/a

**Sponsor Signatory:** 

Ronald Farkas, MD

Chief Medical Officer

25 June 202/

Date

# **Table of Contents**

| 1 | Protocol Summary | 5 |
|-------|-------------------------------------------------------|----|
| 1.1 | Synopsis | 5 |
| 1.2 | Schedule of Activities (SoA) | 7 |
| 2 | Introduction | 8 |
| 2.1 | Study Rationale | 8 |
| 2.2 | Background | 8 |
| 2.2.1 | Obstructive Sleep Apnea | 8 |
| 2.2.2 | Unmet Medical Need | 8 |
| 2.2.3 | Biological Rationale | 9 |
| 3 | Endpoints | 10 |
| 4 | Study Design | 11 |
| 4.1 | Overall Design | 11 |
| 4.2 | Scientific Rationale for Study Design and Dose | 12 |
| 4.3 | End of Study Definition | 13 |
| 5 | Study Population | 13 |
| 5.1 | Inclusion Criteria | 13 |
| 5.2 | Exclusion Criteria | 14 |
| 5.3 | Meals and Dietary Restrictions | 16 |
| 5.4 | Caffeine, Alcohol, and Tobacco | 16 |
| 5.5 | Activity | 17 |
| 5.6 | Screen Failures | 17 |
| 6 | Study Drug | 18 |
| 6.1 | Study Treatment(s) Administered | 18 |
| 6.2 | Preparation/Handling/Storage/Accountability | 18 |
| 6.3 | Concomitant Therapy | 19 |
| 6.4 | Discontinuation of Study Treatment. | 21 |
| 6.5 | Stopping Criteria | 21 |
| 6.5.1 | Individual Participant Stopping Criteria | 21 |
| 6.6 | Participant Discontinuation/Withdrawal from the Study | 21 |
| 6.7 | Loss of Participants to Follow-Up | 22 |
| 7 | Study Assessments and Procedures | 23 |
| 7.1.1 | Polysomnography | 23 |
| 7.2 | Safety Assessments | 23 |

V1.0

| 7.2.1 | Physical Examinations | 24 |
|---|---|---|
| 7.2.2 | Vital Signs | 24 |
| 7.2.3 | Electrocardiograms | 24 |
| 7.2.4 | Clinical Safety Laboratory Assessments | 24 |
| 7.3 | Adverse Events and Serious Adverse Events | 25 |
| 7.3.1 | Time Period and Frequency for Collecting AE and SAE Information | 25 |
| 7.3.2 | Method of Detecting AEs and SAEs | 25 |
| 7.3.3 | Follow-up of AEs and SAEs | 26 |
| 7.3.4 | Regulatory Reporting Requirements for SAEs | 26 |
| 7.3.5 | Pregnancy | 26 |
| 7.4 | Treatment of Overdose | 27 |
| 7.5 | Pharmacokinetics | 27 |
| 8 | Statistical Considerations | 28 |
| 8.1 | Sample Size Determination | 28 |
| 8.2 | Populations for Analyses | 28 |
| 8.3 | Interim Analyses | 28 |
| 9 | Supporting Documentation and Operational Considerations | 28 |
| 9.1 | Appendix 1: Regulatory, Ethical, and Study Oversight Considerations | 28 |
| 9.1.1 | Regulatory and Ethical Considerations | 29 |
| 9.1.2 | Financial Disclosure | 29 |
| 9.1.3 | Informed Consent Process | 30 |
| 9.1.4 | Data Protection | 30 |
| 9.1.5 | Data Quality Assurance | 30 |
| 9.1.6 | Source Documents | 31 |
| 9.1.7 | Study and Site Closure | 31 |
| 9.1.8 | Publication Policy | 32 |
| 9.1.9 | Protocol Approval and Amendment | 32 |
| 9.1.10 | Liability and Insurance | 33 |
| 9.2 | Appendix 2: Clinical Laboratory Tests | 33 |
| 9.3 | Appendix 3: Adverse Events: Definitions and Procedures for Recording, Evaluate Follow-up, and Reporting | • |
| 9.4 | Appendix 4: Contraceptive Guidance and Collection of Pregnancy Information | |
| 9.5 | Appendix 5: List of Abbreviations | 43 |
| 10 | References | 45 |

Apnimed, Inc.

Protocol: SEED

Clinical Study Protocol

### 1 Protocol Summary

### 1.1 Synopsis

**Protocol Title:** Open-Label 4-Period Dose-Escalation Safety and Efficacy Study of AD313 in Participants With Obstructive Sleep Apnea

**Sponsor Study Name.: SEED** 

**Sponsor:** Apnimed, Inc.

#### **Rationale:**

Selective norepinephrine reuptake inhibitors (SNRIs) such as atomoxetine are thought to improve obstructive sleep apnea (OSA) by increasing pharyngeal muscle stiffness and responsiveness.

Cannabinoids, including dronabinol, also have shown potential for reduction of OSA severity. The mechanism of beneficial action of dronabinol appears to be distinct from that of SNRIs, potentially involving stabilization of respiratory patterns and increased activation of upper airway dilating muscles during sleep.

The SEED study is designed to assess the safety and efficacy for OSA of 3 escalating dose combinations of atomoxetine with dronabinol, compared to baseline and to atomoxetine alone.

### **Overall Design:**

The SEED study is an open-label, 4 consecutive period dose-escalation study of combinations of atomoxetine with dronabinol vs. atomoxetine alone in participants with moderate- to severe OSA. A screening polysomnogram (PSG) will be conducted to establish that each participant meets study enrollment criteria and to serve as baseline. Each participant will then receive escalating doses of atomoxetine, then escalating doses of the combination of atomoxetine with dronabinol, as follows:

- Week 1: atomoxetine 40 mg x 3 days, then atomoxetine 80 mg x 4 days
- Week 2: atomoxetine 40 mg/dronabinol 2.5 mg
- Week 3: atomoxetine 80 mg/dronabinol 5 mg
- Week 4: atomoxetine 80 mg/dronabinol 10 mg

25 June 2021 5 of 47 V1.0

Dosing of study drug occurs at the participants usual bedtime. Dose escalation will be based on safety and tolerability, as assessed at weekly clinic visits and telephone contact with participants mid-week of each dosing period.

In addition to the screening/baseline PSG, three on-drug PSGs will be conducted on the final night of the following dosing periods:

- 1<sup>st</sup> week, dosing atomoxetine 80 mg alone
- 3<sup>rd</sup> week, dosing atomoxetine 80 mg/dronabinol 5 mg
- 4<sup>th</sup> week, dosing atomoxetine 80 mg/dronabinol 10 mg

### **Number of Participants:**

A total of 15 participants will be enrolled.

### **Study Duration:**

The overall study duration will be up to 9 weeks, as follows:

- Screening, up to 3 weeks;
- Atomoxetine alone: 1 week
- Dronabinol dose escalation period: 3 weeks
- End of Study telephone contact: 2 weeks

# 1.2 Schedule of Activities (SoA)

Table 1Schedule of Activities

| | | Screening/ | Dosing Period | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Non-PSG<br>Screening<br>V1 | Baseline<br>PSG<br>V2 | ATO 40 3d, ATO 80 4d | | ATO 40/DRO 2.5 | | ATO 80/DRO 5 | | ATO 80/DRO 10 | | |
| Procedures | | | At home<br>dosing | V3<br>PSG | At home dosing | V4 | At home dosing | V5 | At home dosing | PSG<br>V6 | EoS Call |
| Day <sup>1</sup> | -21 t | o -1 | $1 - 7 \pm 1$ | 7 ± 1 | $8-14 \pm 2$ | $14 \pm 2$ | $15 - 21 \pm 2$ | $21 \pm 2$ | $21-28 \pm 2$ | $28 \pm 2$ | 42± 2 |
| Informed consent | X | | | | | | | | | | |
| Demography | X | | | | | | | | | | |
| Physical exam | X | | | | | | | | | | |
| Medical history | X | | | | | | | | | | |
| Pregnancy test <sup>2</sup> | X | | | | | | | | | | |
| Clinical laboratory testing | X | | | | | | | | | | |
| 12 Lead ECG | X | | | | | | | | | | |
| PSG | | $X^3$ | | X | | | | X | | X | |
| Study drug dispense/return | | X | | X | | X | | X | | X | |
| HS study treatment <sup>4</sup> | | | $\leftrightarrow$ | $\leftrightarrow$ | $\leftrightarrow$ | $\leftrightarrow$ | $\leftrightarrow$ | $\leftrightarrow$ | $\leftrightarrow$ | $\leftrightarrow$ | |
| PGI-S, PROMIS sleep<br>impairment, PROMIS sleep<br>disturbance, PROMIS fatigue,<br>DSST, VOLT, PVT <sup>5</sup> | | X | | X | | | | X | | X | |
| Vital signs <sup>6</sup> | X | X | | X | | X | | X | | X | |
| AE/SAE monitoring <sup>7</sup> | | | $\leftrightarrow$ | $\leftrightarrow$ | $\leftrightarrow$ | $\leftrightarrow$ | $\leftrightarrow$ | $\leftrightarrow$ | $\leftrightarrow$ | $\leftrightarrow$ | $\leftrightarrow$ |
| Prior/concomitant medication | | | $\leftrightarrow$ | $\leftrightarrow$ | $\leftrightarrow$ | $\leftrightarrow$ | $\leftrightarrow$ | $\leftrightarrow$ | $\leftrightarrow$ | $\leftrightarrow$ | $\leftrightarrow$ |

Abbreviations: AE = adverse event; ATO = atomoxetine; DRO = dronabinol; DSST = Digit symbol substitution test; ECG = electrocardiogram; HS = Hora Somni; PGI-S = patient global impression of severity of OSA; PSG = polysomnography; SAE = serious adverse event; SAQLI = Sleep Apnea Quality of Life Index; WOCBP = women of childbearing potential; PROMIS = Patient Reported Outcomes Measurement Information System; PVT = psychomotor vigilance test; VOLT = visual object learning task

25 June 2021 7 of 47 V1.0

 $<sup>^{1}</sup>$ Study days shown represent case with no use of  $\pm$  window days; study days shift cumulatively if window days are used

<sup>&</sup>lt;sup>2</sup> WOCBP only

<sup>&</sup>lt;sup>3</sup> On a case-by-case basis with agreement of Sponsor a PSG conducted at the site within 3 months may be used instead of the Screening PSG

<sup>&</sup>lt;sup>4</sup> Study medication administered at lights out; dose on PSG nights is from supply dispensed to the participant if available, but can be provided from separate site supply.

<sup>&</sup>lt;sup>5</sup> Administered at similar time on morning of each PSG visit

<sup>&</sup>lt;sup>6</sup> Vital signs include seated blood pressure in triplicate, pulse, respiratory rate; vital signs on PSG nights taken morning after PSG.

<sup>&</sup>lt;sup>7</sup> Site contacts participant by telephone mid-week of each at-home dosing period for safety evaluation and reminder of study activities

#### 2 Introduction

### 2.1 Study Rationale

Selective norepinephrine reuptake inhibitors (SNRIs) such as atomoxetine are thought to improve obstructive sleep apnea (OSA) by increasing pharyngeal muscle stiffness and responsiveness (1-4).

Cannabinoids, such as dronabinol, have shown potential for reduction of OSA severity (21). The mechanism of beneficial action of dronabinol appears to be distinct from that of SNRIs, potentially involving stabilization of respiratory patterns and increased activation of upper airway dilating muscles during sleep.

The SEED study is designed to assess the safety and efficacy for OSA of 3 escalating dose combinations of atomoxetine and dronabinol.

### 2.2 Background

### 2.2.1 Obstructive Sleep Apnea

The National Commission on Sleep Disorders Research identified sleep disorders as a major public health burden. OSA is the most common and serious of these sleep disorders and affects approximately 20 million people in the United States (US), with approximately 13% of men and 6% of women affected (5). OSA is characterized by repetitive collapse or 'obstruction' of the pharyngeal airway during sleep, manifesting as repetitive episodes of hypopnea (i.e., shallow breathing) or apnea (i.e., paused breathing). These episodes of hypopnea or apnea may lead to arousal from sleep, sleep fragmentation, excessive daytime sleepiness, and/or neuropsychological impairment.

Research has shown that a number of pathogenic factors, or traits, contribute to the development of OSA (6-9). The most important factors are the presence of an anatomically small, collapsible upper airway and a loss of pharyngeal muscle tone or responsiveness during sleep.

Long-term, OSA is associated with increased mortality and a number of adverse cardiovascular, neurocognitive, metabolic, and daytime functioning consequences (10-19).

#### 2.2.2 Unmet Medical Need

Treatment for OSA changed little over the past 40 years, with the overwhelming majority of patients treated with positive airway pressure, the most common of which is continuous positive airway pressure (CPAP), provided by a machine that mechanically maintains an open airway.

Other treatments, such as pharyngeal surgery, mandibular advancement devices, and implantable nerve stimulators, were developed to address the anatomical predisposition to collapse; however, they have shown limited efficacy for niche populations.

While CPAP and related therapies are effective in improving sleep characteristics and oxygenation, many, perhaps most, patients find these devices uncomfortable or intolerable, and most estimates indicate that fewer than 50% of patients prescribed CPAP use it more than 4 hours per night, if at all (20). Efforts to develop pharmacologic therapies, such as antidepressants, stimulants, and hormonal agents, for the treatment of OSA have been ongoing for at least 20 years, with no success thus far.

As many patients cannot use CPAP because they find it intolerable, this represents a significant health concern, as OSA is associated with numerous co-morbidities and increased mortality. Alternative options, such as drugs that activate the pharyngeal muscles, are needed.

### 2.2.3 Biological Rationale

Atomoxetine is a pre-synaptic norepinephrine reuptake inhibitor indicated for the treatment of attention deficit hyperactivity disorder in children and adults. Dronabinol is synthetic delta-9-tetrahydrocannabinol (delta-9-THC) indicated for the treatment of anorexia in patients with AIDS and nausea and vomiting associated with cancer chemotherapy. Apnimed believes that the combination of dronabinol and atomoxetine may have an improved efficacy profile in patients with OSA compared to either constituent alone.

# 3 Endpoints

| | Endpoints |
|---|---|
| Primary | AHI4%, ATO 80/DRO 10 vs. baseline |
| Secondary | <ul> <li>AHI4%, ATO 80/DRO 10 vs. ATO 80</li> <li>AHI4%, ATO 80/DRO 5 vs. baseline</li> <li>AHI4%, ATO 80/DRO 5 vs. ATO 80</li> <li>HB4%, ODI4%, Total time with SaO<sub>2</sub> &lt;90%, Proportion of participants with ≥50% reduction in AHI4%, HB4%, ODI4%</li> </ul> |
| Exploratory | <ul> <li>PGI-S</li> <li>PROMIS sleep impairment</li> <li>PROMIS sleep disturbance</li> <li>PROMIS fatigue</li> <li>AHI4%, highest dose achieved by patient (ie ATO 80/DRO 5 or ATO 80/DRO 10 vs. baseline and vs. ATO 80</li> <li>AHI3 (hypopnea scored when associated with 3% O<sub>2</sub> desaturation)</li> <li>AHI3a (hypopnea scored when associated with 3% O<sub>2</sub> desaturation or arousal)</li> <li>OSA endotype endpoints (Vpassive, Vactive, Muscle Compensation, Loop Gain)</li> <li>PSG sleep and arousal parameters</li> </ul> |
| <b>Safety Endpoints</b> | Vital signs, Spontaneous adverse events, DSST, VOLT, PVT |

Abbreviations: AHI = apnea-hypopnea index; ATO = atomoxetine; DSST = digit symbol substitution test; DRO = dronabinol; HB = hypoxic burden; ODI = Oxygen Desaturation Index; OSA = obstructive sleep apnea; PROMIS = Patient Reported Outcome Measurement Information System; PGI-S = Patient Global Impression of Severity; PSG = polysomnography; PROMIS = Patient Reported Outcome Measurement Information System; PVT = psychomotor vigilance task; SaO<sub>2</sub> = oxygen saturation; SAQLI = Sleep Apnea Quality of Life Index; VOLT = visual object learning task

# 4 Study Design

### 4.1 Overall Design

The SEED study is an open-label, 4 consecutive period dose-escalation study of combinations of atomoxetine and dronabinol in participants with moderate to severe OSA. Participants will undergo initial pre-screening to determine potential study eligibility. Participants selected for further screening should either have a previous history of OSA of a severity consistent with enrollment criteria or be at high risk (e.g. as assessed by STOP-Bang Questionnaire score). Only participants who meet all non-PSG enrollment criteria at Visit 1 are eligible for a screening PSG. On a case by case basis and with agreement of the Sponsor a PSG conducted at the site within 3 months may be used instead of the Screening PSG.

Participants who meet all enrollment criteria will receive an escalating dose of atomoxetine the first week: 3 days of atomoxetine 40 mg followed by 4 days of atomoxetine 80 mg. Participants will then receive escalating dose combinations of atomoxetine and dronabinol for the next 3 weeks. The weekly dose schedule is as follows:

- Week 1: atomoxetine 40 mg x 3 days, then 80 mg x 4 days
- Week 2: atomoxetine 40 mg/dronabinol 2.5 mg
- Week 3: atomoxetine 80 mg/dronabinol 5 mg
- Week 4: atomoxetine 80 mg/dronabinol 10 mg

Dose escalation will be based on safety and tolerability, as assessed at weekly clinic visits and by telephone contact with participants mid-week of each at-home dosing period. Patients who do not tolerate dose escalation will discontinue dosing.

Three on-drug PSGs will be conducted on the final night of the following dosing periods:

- 1st week, dosing atomoxetine 80 mg alone
- 3rd week, dosing atomoxetine 80 mg/dronabinol 5 mg
- 4th week, dosing atomoxetine 80 mg/dronabinol 10 mg

Study drug for Week 1 is dispensed to participants at Visit 2.. Any unused Week 1 study drug is returned at Visit 3. Similarly, study drug for Week 2, 3, and 4 is dispensed at Visits 3, 4 and 5, and unused study drug similarly returned at the subsequent visit.

Dosing of the study treatment will occur each night at the participant's usual bedtime, both during at-home nights and Visit 3, Visit 5 and Visit 6 PSG nights. Study drug dose on PSG nights

is from the supply dispensed to the participant if available, but can be provided from separate site supply.

The morning of each PSG the PGI-S, PROMIS assessments, DSST, VOLT and PVT will be administered.

An End-of-Study phone call will take place 2 weeks following the end of study drug dosing.

Participants who discontinue from the study will not be replaced. No subsequent open-label extension is planned following the study.

Figure 1: Overview of Study Design



EoS = End of Study; PSG = polysomnography; 40 = atomoxetine 40 mg alone; 80 = atomoxetine 80 mg alone; 40/2.5 = atomoxetine 40 mg/dronabinol 2.5 mg; 80/5 = atomoxetine 80 mg/dronabinol 5 mg; 80/10 = atomoxetine 80 mg/dronabinol 10 mg

# 4.2 Scientific Rationale for Study Design and Dose

Selective norepinephrine reuptake inhibitors (SNRIs) such as atomoxetine are thought to improve obstructive sleep apnea (OSA) by increasing pharyngeal muscle stiffness and responsiveness.

Cannabinoids, including dronabinol, also have shown potential for reduction of OSA severity (21). The mechanism of beneficial action of dronabinol appears to be distinct from that of SNRIs, potentially involving stabilization of respiratory patterns and increased activation of upper airway dilating muscles during sleep. Cannabinoids have also shown a hypnotic effect that may counteract the potential wakefulness induced by atomoxetine.

25 June 2021 12 of 47 V1.0

This study is designed to investigate if the combination of atomoxetine and dronabinol is safe and effective in participants with moderate to severe OSA.

### 4.3 End of Study Definition

A participant is considered to have completed the study if he/she has completed all phases of the study through the last scheduled procedure shown in the Schedule of Activities (SoA).

The end of the study is defined as the date of the last visit of the last participant in the study or last scheduled procedure shown in the SoA for the last participant in the study globally.

### 5 Study Population

Eligible participants will be recruited both from the existing clinic population at the study site, including databases of previous subjects who participated in other studies, and through direct advertising to the community.

Participants must be able to provide written consent and meet all the inclusion criteria and none of the exclusion criteria.

#### 5.1 Inclusion Criteria

### Age and Sex

1. 25 to 65 years of age, inclusive, at the Screening Visit.

#### **Disease Measures**

- 2. AHI 10 to 50 (hypopneas defined by 4% oxygen desaturation)
- 3. ≤25% of apneas are central or mixed apneas at V2 baseline PSG

### Weight

4. BMI between 18.5 and 40.0 kg/m<sup>2</sup>, inclusive, at the pre-PSG visit.

### Male participants:

5. If male and sexually active with female partner(s) of childbearing potential, participant must agree, from Study Day 1 through 1 week after the last dose of study drug, to practice

the protocol specified contraception (see Appendix 4: Contraceptive Guidance and Collection of Pregnancy Information).

### Female participants:

- 6. If a woman of childbearing potential (WOCBP), the participant must agree, from Study Day 1 through 1 week after the last dose of study drug, to practice the protocol specified contraception (See Appendix 4: Contraceptive Guidance and Collection of Pregnancy Information). All WOCBP must have negative result of a serum pregnancy test performed at screening.
- 7. If female and of non-childbearing potential, the participant must be either postmenopausal (defined as age ≥ 55 years with no menses for 12 or more months without an alternative medical cause) or permanently surgically sterile (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).

### **Informed Consent**

- 8. Participant voluntarily agrees to participate in this study and signs an Institutional Review Board (IRB)-approved informed consent prior to performing any of the Screening Visit procedures.
- 9. Participant must be able to understand the nature of the study and must have the opportunity to have any questions answered.

### 5.2 Exclusion Criteria

Participants are excluded from the study if any of the following criteria apply:

#### **Medical Conditions**

- 1. History of clinically significant sleep disorder other than OSA.
- 2. Clinically significant craniofacial malformation.
- 3. Clinically significant cardiac disease (e.g., rhythm disturbances, coronary artery disease or cardiac failure) or hypertension requiring more than 2 medications for control (combination medications are considered as 1 medication for this purpose).
- 4. Clinically significant neurological disorder, including epilepsy/convulsions.
- 5. History of schizophrenia, schizoaffective disorder or bipolar disorder according to Diagnostic and Statistical Manual of Mental Disorders-5 (DSM-5) or International Classification of Disease tenth edition criteria.

25 June 2021 14 of 47 V1.0

- 6. History of attempted suicide within 1 year prior to screening, or current suicidal ideation.
- 7. Medically unexplained positive screen for drugs of abuse or history of substance use disorder as defined in DSM-V within 24 months prior to Screening Visit.
- 8. A significant illness or infection requiring medical treatment in the past 30 days.
- 9. Clinically significant cognitive dysfunction as determined by investigator.
- 10. Women who are pregnant or nursing.

### **Prior/Concomitant Therapy**

- 11. History of using devices for OSA treatment, including CPAP, oral or nasal devices, or positional devices, may enroll as long as the devices have not been used for at least 2 weeks prior to first study visit and are not used during participation in the study.
- 12. History of chronic oxygen therapy.
- 13. Use of medications from the list of disallowed concomitant medications.
- 14. Treatment with strong cytochrome P450 3A4 (CYP3A4) inhibitors, strong cytochrome P450 2D6 (CYP2D6) inhibitors, or monoamine oxidase inhibitors (MAOI) within 14 days of the start of treatment, or concomitant with treatment.

### **Prior/Concurrent Clinical Study Experience**

15. Use of another investigational agent within 30 days or 5 half-lives, whichever is longer, prior to dosing.

#### **Diagnostic Assessments**

- 16. Hepatic transaminases >2X the upper limit of normal (ULN), total bilirubin >1.5X ULN (unless confirmed Gilbert syndrome), estimated glomerular filtration rate < 60 ml/min.
- 17. PLM arousal index >20

#### **Other Exclusions**

- 18. <5 hours typical sleep duration.
- 19. ESS > 18
- 20. Night- or shift-work sleep schedule which causes the major sleep period to be during the day.
- 21. Employment as a commercial driver or operator of heavy or hazardous equipment.

25 June 2021 15 of 47 V1.0

- 22. Typically smoking more than 10 cigarettes or 2 cigars per day, or inability to abstain from smoking during overnight PSG visits.
- 23. Unwilling to use specified contraception.
- 24. History of regular alcohol consumption of more than 14 standard units per week (males) or more than 7 standard units per week (females), or unwillingness to limit alcohol consumption to no greater than 2 units/day (males), 1 unit per day (females), not to be consumed within 3 hours of bedtime or on PSG nights.
- 25. Unwilling to limit during the study period caffeinated beverage intake (e.g., coffee, cola, tea) to 400 mg/day or less of caffeine, not to be used within 3 hours of bedtime.
- 26. Any condition that in the investigator's opinion would present an unreasonable risk to the participant, or which would interfere with their participation in the study or confound study interpretation.
- 27. Participant considered by the investigator, for any reason, an unsuitable candidate to receive atomoxetine and/or dronabinol or unable or unlikely to understand or comply with the dosing schedule or study evaluations.

### 5.3 Meals and Dietary Restrictions

- 1. Participants should refrain from consumption of any nutrients known to modulate CYP enzyme activity (e.g., grapefruit or grapefruit juice, pomelo juice, star fruit, pomegranate, and Seville or Moro [blood] orange products) within 72 hours before the first dose of study drug and during the study.
- 2. Diet should be generally stable during the study, e.g., new diet programs should not be initiated.

# 5.4 Caffeine, Alcohol, and Tobacco

- 1. During the outpatient portions of the study, participants should refrain from more than 2 standard units per day of alcohol for men or 1 unit/day for women, consumed no less than 3 hours prior to bedtime. Alcohol should not be consumed on PSG nights.
- 2. Moderate consumption of caffeinated beverages, containing up to a total of 400 mg caffeine per day, is permitted during the study period, consumed no less than 3 hours prior to bedtime.

25 June 2021 16 of 47 V1.0

### 5.5 Activity

There are no restrictions on physical activity during the study other than that physical activity should be generally stable during the study (e.g., new exercise programs should not be initiated).

### 5.6 Screen Failures

Screen failures are defined as participants who consent to participate in the clinical study but are not subsequently assigned to receive study treatment/entered into the study. A minimal set of screen failure information is required to ensure transparent reporting of screen failure participants that meets the Consolidated Standards of Reporting Trials publishing requirements and to respond to queries from regulatory authorities. Minimal information includes demography, screen failure details, eligibility criteria, and any serious adverse events (SAEs).

Individuals who do not meet the criteria for participation in this study (screen failure) will not be rescreened, except if the opportunity for rescreening has been enabled by protocol amendment.

### 6 Study Drug

Study drug is defined as any investigational treatment(s), marketed product(s), placebo, or medical device(s) intended to be administered to a study participant according to the study protocol.

### 6.1 Study Treatment(s) Administered

One capsule of atomoxetine (week 1) or one capsule of atomoxetine and one capsule of dronabinol (weeks 2-4) is taken immediately before the participant's planned bedtime.

| Study Treatment Name: | Atomoxetine hydrochloride | Dronabinol |
|---|---|---|
| <b>Dosage Formulation:</b> | Capsule | Capsule |
| Dosage Levels: | 40 mg, 80 mg | 2.5 mg, 5 mg, 10 mg |
| Route of Administration: | Oral | Oral |
| <b>Dosing Instructions:</b> | 1 capsule administered with up to 240 mL water | 1 capsule administered with up to 240 mL water |
| Storage/Packaging/Labeling: | Store at room temperature, in HDPE bottles | Store at room temperature in HDPE bottles |

# 6.2 Preparation/Handling/Storage/Accountability

- 1. The Investigator or designee must maintain a log to confirm appropriate temperature conditions have been maintained during transit for all study treatments received and any discrepancies are reported and resolved before use of the study treatment.
- 2. Only participants enrolled in the study may receive study treatments and only authorized site staff may supply or administer study treatments. All study treatments must be stored in a secure, environmentally controlled, and monitored (manual or automated) area in accordance with the labeled storage conditions with access limited to the Investigator and authorized site staff.
- 3. The Investigator, institution, or the head of the medical institution (where applicable) is responsible for study treatment accountability, reconciliation, and record maintenance (i.e., receipt, reconciliation, and final disposition records).

4. After receiving Sponsor approval in writing, sites are responsible for returning all unused or partially used study treatment to the Sponsor or designated third party or for preparing the study treatment for destruction via incineration.

# **6.3** Concomitant Therapy

Concomitant therapy with the medications listed below is disallowed. For medication that is typically used as-needed for symptomatic conditions (e.g., occasional use of a sleep aid), the medication should not be used for at least one week prior to the first study PSG and for the duration of the study.

- MAOIs or other drugs that affect monoamine concentrations (e.g., rasagiline) [MAOIs are contraindicated for use with atomoxetine]
- Lithium
- Cannabinoids
- Selective Serotonin Reuptake Inhibitors (e.g., paroxetine)
- Selective Norepinephrine Reuptake Inhibitors (e.g., duloxetine)
- Norepinephrine Reuptake Inhibitors (e.g., reboxetine)
- Alpha-1 antagonists (e.g., tamsulosin)
- Tricyclic antidepressants (e.g., desipramine)
- CYP2D6 inhibitors
- Strong CYP3A4 inhibitors (e.g., ketoconazole)
- Benzodiazepines and other anxiolytics
- Opioids
- Sedatives and sedative-hypnotics, including nonbenzodiazepine "Z-drugs" (zolpidem, zaleplon, eszopiclone)
- Muscle relaxants
- Pressor agents
- Drugs with clinically significant cardiac QT-interval prolonging effects
- Drugs known to lower seizure threshold (e.g., chloroquine)
- Amphetamines

25 June 2021 19 of 47 V1.0

- Antiepileptics
- Antiemetics
- Modafinil or armodafinil
- Beta<sub>2</sub> agonists, (e.g., albuterol)
- Antipsychotics
- Sedating antihistamines
- Pseudoephedrine, phenylephrine, oxymetazoline
- Nicotine replacement products
- Most drugs for Parkinson's, Alzheimer's, Huntington's, Amyotrophic Lateral Sclerosis, or drugs for other neurodegenerative diseases

Medications that do not have substantial effects on the central nervous system (CNS), respiration, or muscle activity are generally allowed including, but not necessarily limited to, the following drugs and drug classes:

- Antihypertensives (angiotensin-converting-enzyme [ACE] /angiotensin II receptor blocker [ARB] inhibitors, calcium channel blockers, hydrochlorothiazide, etc.).
- Statins
- Proton pump inhibitors and histamine h<sub>2</sub> receptor blockers
- Over-the-counter (OTC) antacids
- Non-sedating antihistamines (e.g., cetirizine, loratadine)
- Acetaminophen
- Laxatives
- Erectile dysfunction drugs
- Inhaled corticosteroids (e.g., fluticasone)
- Anti-diabetics
- Ocular hypotensives and other ophthalmics (e.g., timolol)
- Hormonal therapy (e.g., estrogen replacement or anti-estrogens) and hormonal contraceptives

25 June 2021 20 of 47 V1.0

- Thyroid medications
- Anticoagulants
- Osteoporosis drugs

### 6.4 Discontinuation of Study Treatment

If a clinically significant finding is identified, the Investigator or qualified designee will determine if the participant can continue in the study and if any change in participant management is needed. Any new clinically relevant finding should be reported as an adverse event (AE).

# 6.5 Stopping Criteria

### 6.5.1 Individual Participant Stopping Criteria

- Incidents of abuse, diversion, or misuse of the study treatment.
- Incidents of clinical significance: hallucinations, amnesia, delusional thinking, delirium, manic symptoms, aggressive behavior, suicidality, homicidality, agitation, confusion, or convulsions/seizures.
- Participants reporting any SAE considered possibly related or related to study treatment.
- Any other AE that in the judgment of the Investigator necessitates the participant stopping to protect participant safety.

Participants discontinued from dosing will undergo end of study procedures with follow-up monitoring of any AE(s) as clinically indicated.

# 6.6 Participant Discontinuation/Withdrawal from the Study

- A participant may withdraw from the study at any time at his/her own request, or may be withdrawn at any time at the discretion of the Investigator for safety, behavioral, or administrative reasons.
- If the participant withdraws consent for disclosure of future information, the Sponsor may retain and continue to use any data collected before such a withdrawal of consent.
- If a participant withdraws from the study, he/she may request destruction of any samples taken and not tested, and the Investigator must document this in the site study records.

- All participants who withdraw from the study with an ongoing AE must be followed until the
  event is resolved or deemed stable.
- Participation may be terminated before completing the study and the reason recorded as follows:
  - Withdrawal due to AE
  - o Withdrawal due to incident abuse, diversion, or misuse of the study treatment
  - Loss to follow-up
  - Participant withdrew consent at own request
  - o Other

### 6.7 Loss of Participants to Follow-Up

A participant will be considered lost to follow-up if he or she repeatedly fails to return for scheduled visits and is unable to be contacted by the study site. The following actions must be taken if a participant fails to return to the clinic for a required study visit:

- The site must attempt to contact the participant and reschedule the missed visit as soon as possible (and within the visit window, where one is defined) and counsel the participant on the importance of maintaining the assigned visit schedule and ascertain whether or not the participant wishes to and/or should continue in the study.
- In cases in which the participant is deemed lost to follow-up, the Investigator or designee must make every effort to regain contact with the participant (where possible, 3 telephone calls and, if necessary, a certified letter to the participant's last known mailing address or local equivalent methods). These contact attempts should be documented in the participant's medical record/eCRF.
- Should the participant continue to be unreachable, he/she will be considered to have withdrawn from the study.

25 June 2021 22 of 47 V1.0

### 7 Study Assessments and Procedures

- Study procedures and their timing are summarized in the SoA.
- Adherence to the study design requirements, including those specified in the SoA, is essential and required for study conduct.
- All screening evaluations must be completed and reviewed to confirm that potential
  participants meet all eligibility criteria. The Investigator will maintain a screening log to
  record details of all participants screened and to confirm eligibility or record reasons for
  screening failure, as applicable.
- The maximum amount of blood collected from each participant over the duration of the study will not exceed approximately 50 mL.
- Repeat or unscheduled samples may be taken for safety reasons or for technical issues with the samples, as per the Investigator or designee's discretion.

### 7.1.1 Polysomnography

- Methods: Standard overnight PSG recording and data interpretation will be performed in accordance with the American Academy of Sleep Medicine (AASM) scoring manual.
   Participants will be instrumented with standard PSG electrodes. Time of lights out will be established according to the participants' habitual schedule and kept constant across the PSG study nights. The participants will be given 8 hours of time-in bed.
- Participants should be actively encouraged to spend at least 1/3 of the night in the supine position and at least 1/3 of the night in the lateral position on each night of study.

# 7.2 Safety Assessments

- Planned time points for all safety assessments are provided in the SoA.
- Safety monitoring will be guided by the established safety profiles of dronabinol and atomoxetine. Safety assessments will include physical examinations, measurement of vital signs, DSST, VOLT, PVT, monitoring and recording of AEs, SAEs, and pregnancies, recording of study or treatment discontinuations. Effects on OSA and sleep parameters (e.g., sleep time and sleep stages) will also be monitored by PSG.

25 June 2021 23 of 47 V1.0

# 7.2.1 Physical Examinations

- The general physical examination at screening includes an assessment of general appearance and a review of physical systems (dermatologic, head, eyes, ears, nose, mouth/throat/neck, thyroid, lymph nodes, respiratory, cardiovascular, gastrointestinal, extremities, musculoskeletal, neurologic, and psychiatric systems). Height and weight will also be measured and recorded (with shoes removed and wearing light indoor clothing).
- Investigators should pay special attention to clinical signs related to previous serious illnesses.

# 7.2.2 Vital Signs

- Assessment of vital signs (seated blood pressure, pulse rate, body temperature, respiratory rate) will be performed at the time points indicated in the SoA.
- Vital signs will be measured at all visits in a seated position after 5 minutes rest and will
  include temperature, respiratory rate, systolic and diastolic blood pressure, and pulse.
   Measurements should be made in the same arm of the participant at each visit.
- Systolic and diastolic blood pressure will be repeated for a total of 3 measurements, each at least 2 minutes apart.

# 7.2.3 Electrocardiograms

• A 12-lead ECG will be obtained using an ECG machine that automatically calculates the heart rate and measures the PR, QRS, and QT intervals. The ECG will be recorded in the semi-supine position after the participant has rested in this position for at least 10 minutes.

# 7.2.4 Clinical Safety Laboratory Assessments

- Refer to Section 9.2 for the list of screening clinical laboratory tests to be performed and to the SoA for the timing and frequency.
- The Investigator must review the laboratory report and document this review. The laboratory reports must be filed with the source documents.
- All protocol-required laboratory assessments must be conducted in accordance with the laboratory manual and the SoA.

25 June 2021 24 of 47 V1.0

• If laboratory values from laboratory assessments not specified in the protocol and performed at the institution's local laboratory result in the need for a change in participant management or are considered clinically relevant by the Investigator (e.g., are considered to be an SAE or an AE or require dose modification), then the results must be recorded in the eCRF.

#### 7.3 Adverse Events and Serious Adverse Events

The definitions of AEs and SAEs can be found in Appendix 3.Adverse events will be reported by the participant (or, when appropriate, by a caregiver, surrogate, or the participant's legally authorized representative).

The Investigator and any qualified designees are responsible for detecting, documenting, and reporting events that meet the definition of an AE or SAE and remain responsible for following up on AEs that are serious, considered related to the study treatment or the study, or that caused the participant to discontinue the study and/or study treatment.

# 7.3.1 Time Period and Frequency for Collecting AE and SAE Information

All AEs and SAEs will be collected from first dose of study drug until the end of the study at the timepoints specified in the SoA.

All SAEs will be recorded and reported to the Sponsor or designee within 24 hours, as indicated in Appendix 3. The Investigator will submit any updated SAE data to the Sponsor within 24 hours of it being available.

Investigators are not obligated to actively seek AEs or SAEs after the conclusion of study participation. However, if the Investigator learns of any SAE, including a death, at any time after a participant has been discharged from the study, and he/she considers the event to be reasonably related to the study treatment or study participation, the Investigator must promptly notify the Sponsor.

The method of recording, evaluating, and assessing causality of AEs and SAEs and the procedures for completing and transmitting SAE reports are provided in Appendix 3.

# 7.3.2 Method of Detecting AEs and SAEs

Care will be taken not to introduce bias when detecting AEs and/or SAEs. Open-ended and non-leading verbal questioning of the participant is the preferred method to inquire about AE occurrence.

25 June 2021 25 of 47 V1.0

### 7.3.3 Follow-up of AEs and SAEs

After the initial AE/SAE report, the Investigator is required to proactively follow each participant at subsequent visits/contacts. All SAEs will be followed until resolution, stabilization, until the event is otherwise explained, or the participant is lost to follow-up. Further information on follow-up procedures is given in Appendix 3.

### 7.3.4 Regulatory Reporting Requirements for SAEs

- Prompt notification (within 24 hours, see Appendix 3) by the Investigator to the Sponsor of an SAE is essential so that legal obligations and ethical responsibilities towards the safety of participants and the safety of a study treatment under clinical investigation are met.
- The Sponsor has a legal responsibility to notify both the local regulatory authority and other
  regulatory agencies about the safety of a study treatment under clinical investigation. The
  Sponsor will comply with country-specific regulatory requirements relating to safety
  reporting to the regulatory authority, IRB/Independent Ethics Committees (IEC), and
  Investigators.
- Investigator safety reports must be prepared for suspected unexpected serious adverse reactions (SUSAR) according to local regulatory requirements and Sponsor policy and forwarded to Investigators as necessary.
- An Investigator who receives an Investigator safety report describing an SAE or other specific safety information (e.g., summary or listing of SAE) from the Sponsor will file it along with the Investigator's Brochure and will notify the IRB/IEC, if appropriate according to local requirements.

# 7.3.5 Pregnancy

- Details of all pregnancies in female participants after the start of study treatment and until at least 5 terminal half-lives after the last dose will be collected.
- If a pregnancy is reported, the Investigator should inform the Sponsor within 24 hours of learning of the pregnancy and should follow the procedures outlined in Appendix 4.
- Abnormal pregnancy outcomes (e.g., spontaneous abortion, fetal death, stillbirth, congenital anomalies, ectopic pregnancy) are considered to be SAEs.

25 June 2021 26 of 47 V1.0

### 7.4 Treatment of Overdose

For this study, any dose of atomoxetine hydrochloride greater than 80 mg or dronabinol greater than 10 mg more frequently than QHS will be considered an overdose.

In the event of an overdose, the Investigator should refer to the approved product label for advice on overdose and:

- 1. Contact the Medical Monitor immediately.
- 2. Closely monitor the participant for AE/SAE and laboratory abnormalities as medically indicated.
- 3. Obtain a plasma sample for PK analysis within 1 day from the date of the last dose of study treatment if requested by the Medical Monitor (determined on a case- by- case basis).
- 4. Document the quantity of the excess dose as well as the duration of the overdosing in the eCRF.

Decisions regarding dose interruptions or modifications will be made by the Investigator in consultation with the Medical Monitor based on the clinical evaluation of the participant.

### 7.5 Pharmacokinetics

PK parameters are not evaluated in this study.

### 8 Statistical Considerations

# 8.1 Sample Size Determination

In Apnimed studies atomoxetine alone has decreased AHI by 65% or more, and dronabinol has been reported to decrease AHI by about 50% (21). Assuming that 12 participants will complete the trial, the study will have 90% power to detect a treatment difference with baseline at a two-sided 0.05 significance level if the true difference is AHI is 12 units and the within-subject standard deviation 12. Considering an attrition rate of 25%, we will enroll 15 participants to complete the study.

# 8.2 Populations for Analyses

For the purposes of analysis, the following analysis sets are defined:

| Population | Description |
|---|---|
| Enrolled | All participants who signed the ICF (including screening failures). |
| Modified Intent to Treat (mITT) Population | The mITT Population comprises all participants who take at least 1 dose of any of the study treatments, and have at least 1 measurement on the primary endpoint. |
| Safety Population | The Safety Population consists of all participants who receive at least 1 dose of any of the study treatments. Participants will be analyzed for safety based on the treatment received. |
| Per Protocol (PP) Population | The PP Population consists of all participants without any major protocol violations that could influence efficacy assessment. Participants in this population will be analyzed according to the treatment they actually received. |

# 8.3 Interim Analyses

No interim analysis is planned.

# 9 Supporting Documentation and Operational Considerations

# 9.1 Appendix 1: Regulatory, Ethical, and Study Oversight Considerations

### 9.1.1 Regulatory and Ethical Considerations

- This study will be conducted in accordance with the protocol and with:
  - Consensus ethical principles derived from international guidelines including the Declaration of Helsinki and Council for International Organizations of Medical Sciences International Ethical Guidelines.
  - Applicable International Conference on Harmonisation (ICH) Good Clinical Practice (GCP) Guidelines.
  - Applicable laws and regulations.
- The protocol, protocol amendments, ICF, and other relevant documents (e.g., advertisements) must be submitted to an IRB/IEC by the Investigator and reviewed and approved by the IRB/IEC before the study is initiated.
- Any amendments to the protocol will require IEC/IRB approval before implementation of changes made to the study design, except for changes necessary to eliminate an immediate hazard to study participants.
- The Investigator will be responsible for the following:
  - Providing written summaries of the status of the study to the IRB/IEC annually or more frequently in accordance with the requirements, policies, and procedures established by the IRB/IEC.
  - Notifying the IRB/IEC of SAE or other significant safety findings as required by IRB/IEC procedures.
  - Overall conduct of the study at the site and adherence to requirements of 21 Code of Federal Regulations (CFR), ICH GCP guidelines, the IRB/IEC guidelines, European regulation 536/2014 for clinical studies (if applicable), and all other applicable local regulations.

### 9.1.2 Financial Disclosure

Investigators and sub-Investigators will provide the Sponsor with sufficient, accurate financial information in accordance with local regulations to allow the Sponsor to submit complete and accurate financial certification or disclosure statements to the appropriate regulatory authorities. Investigators are responsible for providing information on financial interests during the course of the study and for 1 year after completion of the study.

25 June 2021 29 of 47 V1.0

#### 9.1.3 Informed Consent Process

- The Investigator or his/her representative will explain the nature of the study to the participant or his/her legally authorized representative and answer all questions regarding the study.
- Participants must be informed that their participation is voluntary. Participants will be required
  to sign a statement of informed consent that meets the requirements of 21 CFR 50, local
  regulations, ICH guidelines, Health Insurance Portability and Accountability Act requirements,
  where applicable, and the IRB/IEC or study center.
- The medical record must include a statement that written informed consent was obtained before the participant was enrolled in the study and the date the written consent was obtained. The authorized person obtaining the informed consent must also sign the ICF.
- Participants must be re-consented to the most current version of the ICF(s) during their participation in the study.
- A copy of the signed ICF(s) must be provided to the participant or the participant's legally authorized representative.

If a protocol amendment is required, the ICF may need to be revised to reflect the changes to the protocol. If the ICF is revised, it must be reviewed and approved by the appropriate IEC/IRB, and signed by all participants subsequently enrolled in the study as well as those currently enrolled in the study.

### 9.1.4 Data Protection

- Participants will be assigned a unique identifier by the Sponsor. Any participant records or datasets that are transferred to the Sponsor will contain the identifier only; participant names or any information which would make the participant identifiable will not be transferred.
- The participant must be informed that his/her personal study-related data will be used by the Sponsor in accordance with local data protection law. The level of disclosure must also be explained to the participant.
- The participant must be informed that his/her medical records may be examined by Clinical Quality Assurance auditors or other authorized personnel appointed by the Sponsor, by appropriate IRB/IEC members, and by inspectors from regulatory authorities.

# 9.1.5 Data Quality Assurance

25 June 2021 30 of 47 V1.0

- All participant data relating to the study will be recorded on printed or eCRFs unless
  transmitted to the Sponsor or designee electronically (e.g., laboratory data). The Investigator is
  responsible for verifying that data entries are accurate and correct by physically or
  electronically signing the eCRF.
- The Investigator must maintain accurate documentation (source data) that supports the information entered in the eCRF.
- The Investigator must permit study-related monitoring, audits, IRB/IEC review, and regulatory agency inspections and provide direct access to source data documents.
- The Sponsor or designee is responsible for the data management of this study including quality checking of the data.
- Records and documents, including signed ICF, pertaining to the conduct of this study must be
  retained by the Investigator for 5 years after study completion unless local regulations or
  institutional policies require a longer retention period. No records may be destroyed during the
  retention period without the written approval of the Sponsor. No records may be transferred to
  another location or party without written notification to the Sponsor.
- All data generated by the site personnel will be recorded electronically at each study center using eCRFs. Data from external sources (such as laboratory data) will be entered into the database. Corrections to the data fields will be captured in an audit trail. The reason for change, the name of the person who performed the change, together with the time and date will be logged to provide an audit trail.

#### 9.1.6 Source Documents

- Source documents provide evidence for the existence of the participant and substantiate the integrity of the data collected. Source documents are filed at the Investigator's site.
- Data entered in the eCRF that are transcribed from source documents must be consistent with the source documents or the discrepancies must be explained. The Investigator may need to request previous medical records or transfer records, depending on the study. Also, current medical records must be available.

# 9.1.7 Study and Site Closure

The Sponsor designee reserves the right to close the study site or terminate the study at any time for any reason at the sole discretion of the Sponsor. Study sites will be closed upon study

25 June 2021 31 of 47 V1.0

completion. A study site is considered closed when all required documents and study supplies have been collected and a study site closure visit has been performed.

The Investigator may initiate study site closure at any time, provided there is reasonable cause and sufficient notice is given in advance of the intended termination.

Reasons for the early closure of a study site by the Sponsor or Investigator may include but are not limited to:

- Failure of the Investigator to comply with the protocol, the requirements of the IRB/IEC or local health authorities, the Sponsor's procedures, or GCP guidelines.
- Inadequate recruitment of participants by the Investigator.
- Discontinuation of further study treatment development.

### 9.1.8 Publication Policy

- Authorship will be determined by mutual agreement and in line with International Committee of Medical Journal Editors authorship requirements.
- The Sponsor retains the right to disapprove any submission for publication, including any publication using trial data, including abstracts, presentations or manuscripts.
- A summary of the study results will also be posted in a publicly accessible database (e.g., www.ClinTrials.gov).

# 9.1.9 Protocol Approval and Amendment

Before the start of the study, the study protocol and/or other relevant documents will be approved by the IEC/IRB/Competent Authorities, in accordance with local legal requirements. The Sponsor must ensure that all ethical and legal requirements have been met before the first participant is enrolled in the study.

This protocol is to be followed exactly. To alter the protocol, amendments or exceptions must be written, receive approval from the appropriate personnel, and receive IRB/IEC/Competent Authority approval prior to implementation (if appropriate).

Administrative changes (not affecting the participant benefit/risk ratio) may be made without the need for a formal amendment. All amendments will be distributed to all protocol recipients, with appropriate instructions.

### 9.1.10 Liability and Insurance

The Sponsor will take out reasonable third-party liability insurance cover in accordance with all local legal requirements. The civil liability of the Investigator, the persons instructed by him or her and the hospital, practice, or institute in which they are employed and the liability of the Sponsor with respect to financial loss due to personal injury and other damage that may arise as a result of the carrying out of this study are governed by the applicable law.

The Sponsor will arrange for participants participating in this study to be insured against financial loss due to personal injury caused by the pharmaceutical products being tested or by medical steps taken in the course of the study.

#### 9.1.10.1 Access to Source Data

Regulatory authorities of certain countries, IRBs, IECs, and/or the Sponsor may wish to carry out source data checks and/or on-site audit inspections. Direct access to source data will be required for these inspections and audits; they will be carried out giving due consideration to data protection and medical confidentiality. The Investigator assures the Sponsor of the necessary support at all times.

# 9.2 Appendix 2: Clinical Laboratory Tests

- The tests detailed in Table 2 will be performed by local laboratory.
- Laboratory testing is performed non-fasting.
- Additional tests may be performed at any time during the study as determined necessary by the Investigator or required by local regulations.

**Table 2: Protocol-Required Safety Laboratory Assessments** 

| Laboratory<br>Assessments | Parameters | | |
|---|---|---|---|
| Hematology | Hematocrit Hemoglobin Platelet Count RBC Count | RBC Indices | WBC count with Differential |

| Serum Chemistry | Albumin | ALT |
|---|---|---|
| | BUN | AST |
| | Creatinine | Alkaline phosphatase |
| | Potassium | Calcium |
| | Sodium | Glucose |
| | Bilirubin | Total cholesterol |
| | Total Protein | Chloride |
| | Uric acid | Bicarbonate |
| Other Tests | • Urinalysis | |
| | HbA1c (Screening Visit only) | |
| | • Serum hCG pregnancy test at screening. Additional testing may be performed if needed in WOCBP. | |
| | Urine test of drugs of abuse (marijuana, cocaine, amphetamine, methamphetamine, opiates, phencyclidine) | |

Abbreviations: ALT = alanine aminotransferase; AST = aspartate aminotransferase; BUN = blood urea nitrogen; HbA1c = hemoglobin A1c (glycated hemoglobin); hCG = human chorionic gonadotropin; RBC = red blood cell count; WBC= white blood cell; WOCBP = women of childbearing potential.

Investigators must document their review of each laboratory safety report.

# 9.3 Appendix 3: Adverse Events: Definitions and Procedures for Recording, Evaluating, Follow-up, and Reporting

#### **Definition of AE**

#### **AE Definition**

- An AE is any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the medicinal product.
- NOTE: An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study treatment.

### **Events Meeting the AE Definition**

Any abnormal laboratory test results (hematology, clinical chemistry, or urinalysis) or
other safety assessments (e.g., ECG, radiological scans, vital signs measurements),
including those that worsen from baseline, considered clinically significant in the
medical and scientific judgment of the Investigator (i.e., not related to progression of
underlying disease).

- Exacerbation of a chronic or intermittent pre-existing condition including either an increase in frequency and/or intensity of the condition.
- New conditions detected or diagnosed after study treatment administration even though it may have been present before the start of the study.
- Signs, symptoms, or the clinical sequelae of a suspected drug-drug interaction.
- Signs, symptoms, or the clinical sequelae of a suspected overdose of either study treatment or a concomitant medication. Overdose per se will not be reported as an AE/SAE unless it is an intentional overdose taken with possible suicidal/self-harming intent. Such overdoses should be reported regardless of sequelae.
- "Lack of efficacy" or "failure of expected pharmacological action" per se will not be reported as an AE or SAE. Such instances will be captured in the efficacy assessments. However, the signs, symptoms, and/or clinical sequelae resulting from lack of efficacy will be reported as an AE or SAE if they fulfill the definition of an AE or SAE.

### **Events NOT Meeting the AE Definition**

- Any clinically significant abnormal laboratory findings or other abnormal safety assessments which are associated with the underlying disease, unless judged by the Investigator to be more severe than expected for the participant's condition.
- The disease/disorder being studied or expected progression, signs, or symptoms of the disease/disorder being studied, unless more severe than expected for the participant's condition.
- Medical or surgical procedure (e.g., endoscopy, appendectomy): the condition that leads to the procedure is the AE.
- Situations in which an untoward medical occurrence did not occur (social and/or convenience admission to a hospital).
- Anticipated day-to-day fluctuations of pre-existing disease(s) or condition(s) present or detected at the start of the study that do not worsen.

#### **Definition of SAE**

If an event is not an AE per definition above, then it cannot be an SAE even if serious conditions are met (e.g., hospitalization for signs/symptoms of the disease under study, death due to progression of disease).

| An SAE is defined as any untoward medical occurrence that, at any dose: |
|-------------------------------------------------------------------------|
| Results in death |
| Is life-threatening |

25 June 2021 35 of 47 V1.0

The term 'life-threatening' in the definition of 'serious' refers to an event in which the participant was at risk of death at the time of the event. It does not refer to an event, which hypothetically might have caused death, if it were more severe.

#### Requires inpatient hospitalization or prolongation of existing hospitalization

In general, hospitalization signifies that the participant has been detained (usually involving at least an overnight stay) at the hospital or emergency ward for observation and/or treatment that would not have been appropriate in the physician's office or outpatient setting. Complications that occur during hospitalization are AE. If a complication prolongs hospitalization or fulfills any other serious criteria, the event is serious. When in doubt as to whether "hospitalization" occurred or was necessary, the AE should be considered serious.

Hospitalization for elective treatment of a pre-existing condition that did not worsen from baseline is not considered an AE.

### Results in persistent disability/incapacity

- The term disability means a substantial disruption of a person's ability to conduct normal life functions.
- This definition is not intended to include experiences of relatively minor medical significance such as uncomplicated headache, nausea, vomiting, diarrhea, influenza, and accidental trauma (e.g., sprained ankle) which may interfere with or prevent everyday life functions but do not constitute a substantial disruption.

### Is a congenital anomaly/birth defect

#### Other situations

Medical or scientific judgment should be exercised in deciding whether SAE
reporting is appropriate in other situations such as important medical events that may
not be immediately life-threatening or result in death or hospitalization but may
jeopardize the participant or may require medical or surgical treatment to prevent one
of the other outcomes listed in the above definition. These events should usually be
considered serious.

Examples of such events include invasive or malignant cancers, intensive treatment in an emergency room or at home for allergic bronchospasm, blood dyscrasias, or convulsions that do not result in hospitalization, or development of drug dependency or drug abuse.

### Recording and Follow-up of AE and SAE

#### **AE and SAE Recording**

- When an AE/SAE occurs, it is the responsibility of the Investigator to review all documentation (e.g., hospital progress notes, laboratory, and diagnostics reports) related to the event.
- The Investigator will then record all relevant AE/SAE information in the eCRF.
- It is **not** acceptable for the Investigator to send photocopies of the participant's medical records in lieu of completion of the AE/SAE eCRF page.
- There may be instances when copies of medical records for certain cases are
  requested by the Sponsor. In this case, all participant identifiers, with the exception of
  the participant number, will be blinded on the copies of the medical records before
  submission to the Sponsor.
- The Investigator will attempt to establish a diagnosis of the event based on signs, symptoms, and/or other clinical information. In such cases, the diagnosis (not the individual signs/symptoms) will be documented as the AE/SAE.

### **Assessment of Intensity**

The Investigator will make an assessment of intensity for each AE and SAE reported during the study and assign it to one of the following categories:

- Mild: An event that is easily tolerated by the participant, causing minimal discomfort and not interfering with everyday activities.
- Moderate: An event that causes sufficient discomfort and interferes with normal everyday activities.
- Severe: An event that prevents normal everyday activities. An AE that is assessed as severe should not be confused with an SAE. Severe is a category utilized for rating the intensity of an event; and both AE and SAE can be assessed as severe.

An event is defined as 'serious' when it meets at least one of the predefined outcomes as described in the definition of an SAE, NOT when it is rated as severe.

### **Assessment of Causality**

- The Investigator is obligated to assess the relationship between study treatment and each occurrence of each AE/SAE.
- A "reasonable possibility" of a relationship conveys that there are facts, evidence, and/or arguments to suggest a causal relationship, rather than a relationship cannot be ruled out.
- The Investigator will use clinical judgment to determine the relationship.
- Alternative causes, such as underlying disease(s), concomitant therapy, and other risk factors, as well as the temporal relationship of the event to study treatment administration will be considered and investigated.
- The Investigator will also consult the Investigator's Brochure and/or Product Information, for marketed products, in his/her assessment.
- For each AE/SAE, the Investigator <u>must</u> document in the medical notes that he/she has reviewed the AE/SAE and has provided an assessment of causality.
- There may be situations in which an SAE has occurred and the Investigator has minimal information to include in the initial report to the Sponsor. However, it is very important that the Investigator always make an assessment of causality for every event before the initial transmission of the SAE data to the Sponsor.
- The Investigator may change his/her opinion of causality in light of follow-up information and send an SAE follow-up report with the updated causality assessment.
- The causality assessment is one of the criteria used when determining regulatory reporting requirements.

### Follow-up of AE and SAE

- The Investigator is obligated to perform or arrange for the conduct of supplemental measurements and/or evaluations as medically indicated or as requested by the Sponsor to elucidate the nature and/or causality of the AE or SAE as fully as possible. This may include additional laboratory tests or investigations, histopathological examinations, or consultation with other health care professionals.
- If a participant dies during participation in the study, the Investigator will provide the Sponsor with a copy of any post-mortem findings including histopathology.

25 June 2021 38 of 47 V1.0

- New or updated information will be recorded in the originally completed eCRF.
- The Investigator will submit any updated SAE data to the Sponsor within 24 hours of receipt of the information.

### **Reporting of SAE to Sponsor**

### **SAE Reporting to Sponsor**

- The Investigator must report any SAEs to the Sponsor within 24 hours of becoming aware of the event.
- When calling to report an SAE, state that you are reporting an SAE and give the Investigator's name, your name, the telephone number where you can be reached, and the protocol number and title.
- The Investigator and the Sponsor will review each SAE report and the Sponsor will evaluate the seriousness and the causal relationship of the event to study treatment. In addition, the Sponsor will evaluate the expectedness according to the reference documents (Investigator's Brochure or US product labeling for atomoxetine or dronabinol). Based on the Investigator and Sponsor's assessment of the event, a decision will be made concerning the need for further action.
- After the study is completed at a given site, the electronic data collection tool will be taken off-line to prevent the entry of new data or changes to existing data.
- If a site receives a report of a new SAE from a study participant or receives updated data on a previously reported SAE after the electronic data collection tool has been taken off-line, then the site can report this information on a paper SAE form or by telephone.

All SAEs will be recorded from signing of informed consent until the end of the study. Serious adverse events occurring after the end of the study and coming to the attention of the Investigator must be reported only if they are considered (in the opinion of the Investigator) causally-related to study treatment.

25 June 2021 39 of 47 V1.0

### **Suspected Unexpected Serious Adverse Reactions (SUSARs)**

Any AE that is serious, associated with the use of the study treatment, and unexpected (SUSAR) has additional reporting requirements, as described below.

- If the SUSAR is fatal or life-threatening, associated with study treatment, and unexpected, regulatory authorities and IECs will be notified within 7 calendar days after the Sponsor learns of the event. Additional follow-up (cause of death, autopsy report, and hospital report) information should be reported within an additional 8 days (15 days total).
- If the SUSAR is not fatal or life-threatening but is otherwise serious, associated with study treatment, and unexpected, regulatory authorities and IECs will be notified within 15 calendar days after the Sponsor learns of the event.

The Sponsor will notify the Investigators in a timely fashion of relevant information about SUSARs that could adversely affect the safety of participants. Follow-up information may be submitted if necessary.

The Sponsor will also provide annual safety updates to the regulatory authorities and IECs responsible for the study. These updates will include information on SUSARs and other relevant safety findings.

# 9.4 Appendix 4: Contraceptive Guidance and Collection of Pregnancy Information

#### **Definitions**

#### **WOCBP**

A woman is considered fertile following menarche and until becoming post-menopausal unless permanently sterile (see below).

Women in the following categories are not considered WOCBP:

- 1. Premenarchal
- 2. Premenopausal female with one of the following:
  - Documented hysterectomy
  - Documented bilateral salpingectomy

Documented bilateral oophorectomy

NOTE: Documentation can come from the site personnel's review of the participant's medical records, medical examination, or medical history interview.

### 3. Post-menopausal female

- A post-menopausal state is defined as no menses for 12 months without an alternative medical cause. A high follicle-stimulating hormone (FSH) level in the post-menopausal range may be used to confirm a post-menopausal state in women not using hormonal contraception or hormonal replacement therapy (HRT). However, in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient.
- Females on HRT and whose menopausal status is in doubt will be required to use one of the non-estrogen hormonal highly effective contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status before study enrollment.

### **Contraception Guidance:**

### **Male Participants:**

Male participants with female partners of childbearing potential are eligible to participate if the agree to ONE of the following during the protocol-defined time frame:

- Are abstinent from penile-vaginal intercourse as their usual and preferred lifestyle (abstinent on a long-term and persistent basis) and agree to remain abstinent.
- Agree to use a contraceptive method with a failure rate of <1% per year as described in the table below when having penile-vaginal intercourse with a WOCBP who is not currently pregnant.

In addition, male participants must refrain from donating sperm for the duration of the study and for 3 months after the last dose of study treatment.

Male participants with a pregnant or breastfeeding partner must agree to remain abstinent from penile-vaginal intercourse or to use a male condom during each episode of penile penetration during the protocol-defined time frame.

### **Female Participants**

25 June 2021 41 of 47 V1.0

Female participants of childbearing potential are eligible to participate if they agree to use a highly effective method of contraception consistently and correctly as described in the table below.

### Highly Effective Contraceptive Methods That Are User Dependent<sup>1</sup>

Failure rate of <1% per year when used consistently and correctly.

Combined (estrogen- and progestin-containing) hormonal contraception associated with inhibition of ovulation<sup>2</sup>

- Oral
- Intravaginal
- Transdermal

Progestogen-only hormonal contraception associated with inhibition of ovulation

- Oral
- Injectable

### Highly Effective Contraceptive Methods That Are User Independent<sup>1</sup>

Implantable progestogen-only hormonal contraception associated with inhibition of ovulation

- IUD
- Intrauterine hormone-releasing system (IUS)
- Bilateral tubal occlusion

#### Vasectomized partner

A vasectomized partner is a highly effective contraception method provided that the partner is the sole male sexual partner of the WOCBP and the absence of sperm has been confirmed. If not, an additional highly effective method of contraception should be used.

#### Sexual abstinence

Sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatment. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the study and the preferred and usual lifestyle of the participant.

#### NOTES:

1 Typical use failure rates may differ from those when used consistently and correctly. Use should be consistent with local regulations regarding the use of contraceptive methods for participants participating in clinical studies.

#### **Pregnancy Testing**

25 June 2021 42 of 47 V1.0

- WOCBP should only be included after a confirmed menstrual period and a negative highly sensitive serum pregnancy test.
- Pregnancy testing will be performed whenever a menstrual cycle is missed or when pregnancy is otherwise suspected.

### **Collection of Pregnancy Information:**

### Female participants who become pregnant

- The Investigator will collect pregnancy information on any female participant who becomes pregnant while participating in this study. Information will be recorded on the appropriate form and submitted to the Sponsor within 24 hours of learning of a participant's pregnancy. The participant will be followed to determine the outcome of the pregnancy. The Investigator will collect any follow up information on the participant and the neonate and the information will be forwarded to the Sponsor. Generally, follow up will not be required for longer than 6 to 8 weeks beyond the estimated delivery date. Any termination of the pregnancy will be reported, regardless of fetal state (presence or absence of anomalies) or indication for the procedure.
- While pregnancy itself is not considered to be an AE or SAE, any pregnancy complication or elective termination of a pregnancy will be reported as an AE or SAE. A spontaneous abortion is always considered to be an SAE and will be reported as such. Any post-study pregnancy-related SAE considered reasonably related to the study treatment by the Investigator will be reported to the Sponsor. While the Investigator is not obligated to actively seek this information in former study participants, he or she may learn of an SAE through spontaneous reporting.
- Any female participant who becomes pregnant while participating in the study will be withdrawn from the study.

# 9.5 Appendix 5: List of Abbreviations

AHI apnea-hypopnea index

AE adverse event

Bang Body mass index, Age, Neck circumference, and Gender criteria

BMI body mass index

CFR Code of Federal Regulations

CNS central nervous system

CPAP continuous positive air pressure

CYP2D6 cytochrome P450 2D6

25 June 2021 43 of 47 V1.0

CYP3A4 cytochrome P450 3A4

DSM-5 Diagnostic and Statistical Manual of Mental Disorders, 5th edition

DSST Digit symbol substitution test

ECG electrocardiogram
EEG electroencephalogram

eCRF electronic case report form(s)

EDC electronic data capture

EOS end of study

FSH follicle-stimulating hormone

GCP Good Clinical Practice

HB hypoxic burden

HRT hormone replacement therapy

ICF informed consent form

ICH International Conference on Harmonisation

IEC Independent Ethics CommitteeIRB Institutional Review BoardOSA obstructive sleep apnea

OTC over-the-counter

MAOI monoamine oxidase inhibitor

PK pharmacokinetic(s) PSG polysomnography

PVT Psychomotor vigilance test
OHS 1 dose every night at bedtime

SAE serious adverse event
SAP Statistical Analysis Plan
SoA Schedule of Activities

STOP Snoring, Tiredness, Observed apnea, and Blood pressure criteria

SUSAR suspected unexpected serious adverse reaction

ULN upper limit of normal

US United States

VOLT Visual object learning task

WOCBP woman of childbearing potential

### 10 References

- 1. Taranto-Montemurro L, Messineo L, Azarbarzin A, Vena D, Hess L, Calianese N, et al. Effects of the Combination of Atomoxetine and Oxybutynin on Obstructive Sleep Apnea Endotypic Traits. CHEST. 2020.
- 2. Taranto-Montemurro L, Messineo L, Sands SA, Azarbarzin A, Marques M, Edwards BA, et al. The Combination of Atomoxetine and Oxybutynin Greatly Reduces Obstructive Sleep Apnea Severity. A Randomized, Placebo-controlled, Double-Blind Crossover Trial. American journal of respiratory and critical care medicine. 2019;199(10):1267-76.
- 3. Taranto-Montemurro L, Messineo L, Wellman A. Targeting Endotypic Traits with Medications for the Pharmacological Treatment of Obstructive Sleep Apnea. A Review of the Current Literature. J Clin Med. 2019;8(11).
- 4. Taranto-Montemurro L, Sands SA, Edwards BA, Azarbarzin A, Marques M, de Melo C, et al. Desipramine improves upper airway collapsibility and reduces OSA severity in patients with minimal muscle compensation. The European respiratory journal. 2016;48(5):1340-50.
- 5. Peppard PE, Young T, Barnet JH, Palta M, Hagen EW, Hla KM. Increased prevalence of sleep-disordered breathing in adults. Am J Epidemiol. 2013;177(9):1006-14.
- 6. Eckert DJ, White DP, Jordan AS, Malhotra A, Wellman A. Defining phenotypic causes of obstructive sleep apnea. Identification of novel therapeutic targets. American journal of respiratory and critical care medicine. 2013;188(8):996-1004.
- 7. Wellman A, Eckert DJ, Jordan AS, Edwards BA, Passaglia CL, Jackson AC, et al. A method for measuring and modeling the physiological traits causing obstructive sleep apnea. J Appl Physiol. 2011;110(6):1627-37.
- 8. Younes M. Contributions of upper airway mechanics and control mechanisms to severity of obstructive apnea. American journal of respiratory and critical care medicine. 2003;168(6):645-58.
- 9. Younes M. Role of arousals in the pathogenesis of obstructive sleep apnea. American journal of respiratory and critical care medicine. 2004;169(5):623-33.
- 10. Somers VK, Dyken ME, Clary MP, Abboud FM. Sympathetic neural mechanisms in obstructive sleep apnea. J Clin Invest. 1995;96(4):1897-904.
- 11. Nieto FJ, Young TB, Lind BK, Shahar E, Samet JM, Redline S, et al. Association of sleep-disordered breathing, sleep apnea, and hypertension in a large community-based study. Sleep Heart Health Study. JAMA. 2000;283(14):1829-36.
- 12. Brooks D, Horner RL, Kozar LF, Render-Teixeira CL, Phillipson EA. Obstructive sleep apnea as a cause of systemic hypertension. Evidence from a canine model. J Clin Invest. 1997;99(1):106-9.
- 13. Peppard PE, Young T, Palta M, Skatrud J. Prospective study of the association between sleep-disordered breathing and hypertension. N Engl J Med. 2000;342(19):1378-84.
- 14. Hung J, Whitford EG, Parsons RW, Hillman DR. Association of sleep apnoea with myocardial infarction in men. Lancet. 1990;336(8710):261-4.
- 15. Wessendorf TE, Teschler H, Wang YM, Konietzko N, Thilmann AF. Sleep-disordered breathing among patients with first-ever stroke. J Neurol. 2000;247(1):41-7.
- 16. Hoffstein V. Blood pressure, snoring, obesity, and nocturnal hypoxaemia. Lancet. 1994;344(8923):643-5.

25 June 2021 45 of 47 V1.0

- 17. Shahar E, Whitney CW, Redline S, Lee ET, Newman AB, Nieto FJ, et al. Sleep-disordered breathing and cardiovascular disease: cross-sectional results of the Sleep Heart Health Study. American journal of respiratory and critical care medicine. 2001;163(1):19-25.
- 18. Redline S, Strauss ME, Adams N, Winters M, Roebuck T, Spry K, et al. Neuropsychological function in mild sleep-disordered breathing. Sleep. 1997;20(2):160-7.
- 19. Findley LJ, Unverzagt ME, Suratt PM. Automobile accidents involving patients with obstructive sleep apnea. The American review of respiratory disease. 1988;138(2):337-40.
- 20. Sawyer AM, Gooneratne NS, Marcus CL, Ofer D, Richards KC, Weaver TE. A systematic review of CPAP adherence across age groups: clinical and empiric insights for developing CPAP adherence interventions. Sleep Med Rev. 2011;15(6):343-56.
- 21. Carley DW et al. Pharmacotherapy of apnea by cannabimimetic enhancement, the PACE clinical trial: effects of dronabinol in obstructive sleep apnea. SLEEP. 2018;41(1):1-13

25 June 2021 46 of 47 V1.0

Apnimed, Inc.

Protocol: SEED

Clinical Study Protocol

### **Declaration of the Investigator**

**Title:** Open-Label 4-Period Dose-Escalation Safety and Efficacy Study of AD313 in Participants With Obstructive Sleep Apnea

All documentation for this study that is supplied to me and that has not been previously published will be kept in the strictest confidence. This documentation includes this study protocol, Investigator's Brochure, EDC system/eCRF, and other scientific data.

The study will not be commenced without the prior written approval of a properly constituted IRB or IEC. No changes will be made to the study protocol without the prior written approval of the Sponsor and the IRB or IEC, except where necessary to eliminate an immediate hazard to the participants.

I have read and understood and agree to abide by all the conditions and instructions contained in this protocol.

# Responsible Investigator of the local study center

| Signature | Date |
|-----------------------------|------|
| Name (block letters) | |
| Title (block letters) | |
| Institution (block letters) | |
| Phone number | |